CLINICAL TRIAL: NCT04272554
Title: Screening/Observational Protocol to Determine Patient Eligibility for Inclusion in AAV Gene Therapy Clinical Trials (ECLIPSE)
Brief Title: AAV Gene Therapy Screening/Observational Protocol (ECLIPSE)
Acronym: ECLIPSE
Status: Completed | Type: Observational
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: FLT-01
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Hemophilia B; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorder; Haematologic Disease
MeSH Terms: conditions — Hemophilia B; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: None Retained — Pharmacogenomic and research biomarker samples will be collected from consenting patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Freeline is developing adeno-associated virus (AAV) vector based gene therapies for a number of diseases and is actively advancing a programme in Haemophilia B (HB). This study aims to collect prospective data to characterise bleeding events and Factor IX (FIX) concentrate consumption in HB patients that can be used as baseline for participants who elect to participate in a subsequent Freeline gene therapy study. The study will also screen participants for antibodies to a novel AAV vector to assess their suitability for inclusion in a Freeline gene therapy treatment study.

DETAILED DESCRIPTION:
This is a prospective study to collect baseline disease characteristics in patients with HB that are required to establish eligibility for treatment with a novel AAV gene therapy in a subsequent Freeline gene therapy treatment study.

Participants providing consent will attend an enrolment visit to complete eligibility evaluations, collect health and demographic information and receive instruction for completing the study diary. Participants will then complete a diary recording bleeding episodes and FIX usage until they enrol into a gene therapy treatment study. A blood sample will be drawn at a convenient timepoint during the study to assess the participant's AAV neutralising antibody (NAb) status.

No treatment intervention will occur as part of this study.

ELIGIBILITY:
Inclusion Criteria

1. Male participants, ≥ 16 years of age.
2. Able to give full informed consent or obtain full informed consent/assent (according to local regulations) and/or obtain full informed consent from the participant's legally acceptable representative (as appropriate), and able to understand and comply with all requirements of the study, including diary completion.
3. Interested in participation in future gene therapy clinical studies.
4. Subjects with Haemophilia B with known severe or moderately severe FIX deficiency (≤2% of normal circulating FIX activity) for which the subject is either on

   1. Continuous routine FIX prophylaxis, OR
   2. On demand FIX treatment
5. If receiving prophylaxis, participant has been on stable and adequate prophylaxis for at least 2 months prior to enrolment.

Exclusion Criteria:

1. Documented evidence of liver fibrosis and/ or liver dysfunction
2. Prior treatment with a gene transfer medicinal product.
3. Known presence or history of neutralising anti-human FIX antibodies (inhibitors)
4. Previously established serological evidence of HIV-1
5. Documented active hepatitis B or C, and HBsAg or HCV RNA viral load positivity, respectively, or currently on antiviral therapy for hepatitis B or C
6. Participants at high risk of thromboembolic events (history of arterial or venous thromboembolism
7. Known coagulation disorder other than Haemophilia B
8. Known history of an allergic reaction or anaphylaxis to Factor IX products or known uncontrolled allergic conditions
9. Known history of allergy to corticosteroids or to tacrolimus or any other macrolide
10. Known medical condition that would require chronic administration of corticosteroids (excluding topical formulations)
11. History of alcohol or drug dependence.
12. Planned surgical procedure within the next 12 months requiring prophylactic FIX treatment.
13. Known active severe infection (including documented COVID-19 infection), or any other significant concurrent, uncontrolled medical condition evaluated by the investigator to interfere with adherence to the protocol procedures or with tolerance to gene therapy in a future treatment study including, but not limited to, renal, hepatic, cardiovascular, opthalmological, hematological, immunological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease, malignancy or any other psychological disorder.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophila B patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Bleeding episodes | 6 - 24 months
  Bleeding episode data recorded during the study
Factor IX replacement therapy consumption | 6 - 24 months
  Factor IX replacement therapy data recorded during the study

SECONDARY OUTCOMES:
To screen Haemophilia B patients for neutralising antibodies to a novel AAV vector (AAVS3). | 6 - 24 months
  AAV antibody assay result
To characterise baseline clinical parameters related to Haemophilia B. | 6 - 24 months
  Target joint data and health reasource utilisation

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, Dr, Principal Investigator — The Royal Free Hospital
Locations (56):
- United States (17):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California - Davis, Sacramento, California
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hemophilia Center of Western New York, Buffalo, New York
  - University of North Carolina (UNC), Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Lombardi Comprehensive Cancer Center at Georgetown University, Georgetown, Washington
  - Blood Center of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Children's Hospital, Parkville, Melbourne
  - The Alfred Hospital, Melbourne
  - Calvary Mater Hospital, Newcastle
  - Royal Prince Alfred Hospital, Sydney
  - Westmead Hospital, Sydney
- Medical University of Vienna, Vienna, Austria
- Canada (5):
  - McMaster University Medical Centre, Hamilton
  - Lawson Health Research Institute, London
  - The Moncton Hospital, Moncton
  - Saskatoon City Hospital, Saskatoon
  - University of Alberta Hospital, Winnipeg
- France (3):
  - Hôpital Louis Pradel - HCL, Bron
  - CHU Bicetre, Paris
  - Hopital Necker-Enfants Malades - AP-HP, Paris
- Germany (2):
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
  - Universitaetsklinikum des Saarlandes und Medizinische Fakultaet der Universitaet des Saarlandes, Homburg
- St James Hospital, Dublin, Ireland
- Italy (4):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Citta della Salute e della Scienza di Torino - Ospedale le Molinette, Torino
- Netherlands (3):
  - Groningen UMC, Groningen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- South Africa (2):
  - University of Cape Town Clinical Research Center, Cape Town
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
- Turkey (Türkiye) (4):
  - Istanbul University Faculty of Medicine, Istanbul
  - Ege University Medical Faculty, Izmir
  - Samsun Ondokuz Mayis University Medical Faculty, Samsun
  - Özel Acibadem Adana Hastanesi, Seyhan
- United Kingdom (9):
  - The Haemophilia and Thrombosis Centre, Canterbury, Kent
  - Queen Elizabeth Hospital, Birmingham
  - Cardiff University Hospital, Cardiff
  - Glasgow Royal Infirmary, Glasgow
  - Hammersmith Hospital, London
  - Royal Free London NHS Foundation Tust, London
  - St Thomas' Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Newcastle Hemophilia Comprehensive Care Centre, Newcastle

IPD SHARING:
Plan to Share IPD: No